CLINICAL TRIAL: NCT02831712
Title: Effect of Iron Status on Occurrence of Non-transferrin-bound Iron (NTBI) in Serum in Response to an Oral Iron Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Walczyk (Other)
Responsible Party: Sponsor-Investigator, Thomas Walczyk, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13-093
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Effect of Iron Status on Occurrence of NTBI
Keywords: NTBI; Iron status; Iron supplement
MeSH Terms: interventions — ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron supplement (Other): Ferrous Fumarate tablet 200 mg
  Interventions: Dietary Supplement: Ferrous Fumarate

INTERVENTIONS:
Dietary Supplement: Ferrous Fumarate — One tablet of a commercial iron supplement (Ferrous Fumarate 200 mg, from Drug House of Australia) will be provided to participants after overnight fast. The intervention is only one time.

SUMMARY:
This study aims to investigate a possible effect of iron status on temporary build-up of non-transferrin bound iron (NTBI) in healthy volunteers upon iron supplementation.

DETAILED DESCRIPTION:
For Visit 1, blood samples will be collected to assess iron status. For Visit 2, after an overnight fast, iron supplement will be provided to participant before breakfast. Blood samples will be collected right before and 2 h after iron supplement consumption for NTBI analysis.

NTBI concentration before and after iron supplement consumption will be compared. Dependence of NTBI formation on markers of iron status (serum iron, transferrin, transferrin saturation, serum ferritin and hemoglobin) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers (21 - 55 years old)
* C-reactive protein (CRP) < 5

Exclusion Criteria:

* Blood donation or significant blood loss (e.g. surgery) within the past 4 months
* Regular intake of iron and other nutrient supplements within the past 4 months
* Regular intake of medication except oral contraceptives
* Acute or recent inflammatory or infectious symptoms
* Chronic gastrointestinal disorders or metabolic diseases
* Pregnancy or lactation
* Coeliac disease or gluten-related disorders
* Iron overload conditions (serum ferritin concentration > 200 ng/mL for females, > 300 ng/mL for males)
* Non iron deficiency anemia [serum ferritin concentration within normal range (15-200 ng/mL for females, 30-300 ng/mL for males) but low hemoglobin (< 12 g/dL for females, < 14 g/dL for males)]

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of NTBI after an oral iron load | 2 hour post dose
  Blood samples collected 2 h after the iron supplement consumption will be measured for NTBI concentration

SECONDARY OUTCOMES:
Dependence of NTBI concentration on markers of iron status (concentrations of serum iron, serum ferritin, transferrin saturation) | 2 hour post dose
  Correlation between NTBI concentration and iron status indicators will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walczyk, Ph.D, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore; National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Malyszko J, Glowinska I, Malyszko JS, Levin-Iaina N, Koc-Zorawska E, Mysliwiec M. Iron metabolism in kidney allograft recipients: still a mystery? Transplant Proc. 2011 Oct;43(8):2973-5. doi: 10.1016/j.transproceed.2011.08.055. PMID 21996204
- [Background] Inati A, Musallam KM, Cappellini MD, Duca L, Taher AT. Nontransferrin-bound iron in transfused patients with sickle cell disease. Int J Lab Hematol. 2011 Apr;33(2):133-7. doi: 10.1111/j.1751-553X.2010.01224.x. PMID 21382180
- [Background] Ounjaijean S, Westermarck T, Partinen M, Plonka-Poltorak E, Kaipainen P, Kaski M, Fucharoen S, Srichairatanakool S, Atroshi F. Increase in non-transferrin bound iron and the oxidative stress status in epilepsy patients treated using valproic acid monotherapy. Int J Clin Pharmacol Ther. 2011 Apr;49(4):268-76. doi: 10.5414/CP201466. PMID 21429441
- [Background] Prakash M, Upadhya S, Prabhu R. Serum non-transferrin bound iron in hemodialysis patients not receiving intravenous iron. Clin Chim Acta. 2005 Oct;360(1-2):194-8. doi: 10.1016/j.cccn.2005.04.024. PMID 15979061
- [Background] Yegin ZA, Pasaoglu H, Aki SZ, Ozkurt ZN, Demirtas C, Yagci M, Acar K, Sucak GT. Pro-oxidative/antioxidative imbalance: a key indicator of adverse outcome in hematopoietic stem cell transplantation. Int J Lab Hematol. 2011 Aug;33(4):414-23. doi: 10.1111/j.1751-553X.2011.01297.x. Epub 2011 Feb 10. PMID 21310008
- [Background] Duca L, Da Ponte A, Cozzi M, Carbone A, Pomati M, Nava I, Cappellini MD, Fiorelli G. Changes in erythropoiesis, iron metabolism and oxidative stress after half-marathon. Intern Emerg Med. 2006;1(1):30-4. doi: 10.1007/BF02934717. PMID 16941810
- [Background] Trumbo P, Yates AA, Schlicker S, Poos M. Dietary reference intakes: vitamin A, vitamin K, arsenic, boron, chromium, copper, iodine, iron, manganese, molybdenum, nickel, silicon, vanadium, and zinc. J Am Diet Assoc. 2001 Mar;101(3):294-301. doi: 10.1016/S0002-8223(01)00078-5. No abstract available. PMID 11269606
- [Background] Monsen ER, Hallberg L, Layrisse M, Hegsted DM, Cook JD, Mertz W, Finch CA. Estimation of available dietary iron. Am J Clin Nutr. 1978 Jan;31(1):134-41. doi: 10.1093/ajcn/31.1.134. PMID 619599
- [Background] Papanikolaou G, Pantopoulos K. Iron metabolism and toxicity. Toxicol Appl Pharmacol. 2005 Jan 15;202(2):199-211. doi: 10.1016/j.taap.2004.06.021. PMID 15629195
- [Background] Hutchinson C, Al-Ashgar W, Liu DY, Hider RC, Powell JJ, Geissler CA. Oral ferrous sulphate leads to a marked increase in pro-oxidant nontransferrin-bound iron. Eur J Clin Invest. 2004 Nov;34(11):782-4. doi: 10.1111/j.1365-2362.2004.01416.x. No abstract available. PMID 15530152
- [Background] Baron J, Ben-David G, Hallak M. Changes in non-transferrin-bound iron (NTBI) in pregnant women on iron supplements. Eur J Obstet Gynecol Reprod Biol. 2008 Oct;140(2):281-2. doi: 10.1016/j.ejogrb.2008.01.002. Epub 2008 Mar 4. No abstract available. PMID 18304722
- [Background] Schumann K, Kroll S, Romero-Abal ME, Georgiou NA, Marx JJ, Weiss G, Solomons NW. Impact of oral iron challenges on circulating non-transferrin-bound iron in healthy Guatemalan males. Ann Nutr Metab. 2012;60(2):98-107. doi: 10.1159/000336177. Epub 2012 Mar 6. PMID 22398912